CLINICAL TRIAL: NCT05564468
Title: Testing the Utility of a Novel Website to Help Cancer Patients Plan for Their Future - Phase 2
Brief Title: Design and Testing of a Web-Based Tool for the Improvement of End-of-Life Planning in Patients With Advanced Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Peacefully, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RG1123556; R44NR020341 (NIH); NCI-2024-03279 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20230 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Locally Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Peacefully's) (Experimental): Patients receive Peacefully's web-based tool to help with end-of-life planning on day 7.
  Interventions: Other: Internet-Based Intervention; Other: Questionnaire Administration
- Group II (standard of care) (Active Comparator): Patients receive standard care.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: Group II (standard of care)
Other: Internet-Based Intervention — Receive Peacefully's end-of-life planning program
  Arms: Group I (Peacefully's)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial examines a web-based tool, in partnership with Peacefully, Inc, designed to improve end-of-life planning among patients with advanced cancers. This program helps users prepare comprehensively for end-of-life (e.g., medical wishes, legal estate planning, financial planning and transfer of accounts, legacy building, and emotional support). It is expected that this web-based end-of-life planning program may reduce distress and improve end-of-life preparation among advanced cancer patients.

DETAILED DESCRIPTION:
OUTLINE:

Patients are randomized to 1 of 2 groups and their engagement in end-of-life planning is assessed at baseline and four weeks post-randomization.

Group I (intervention): Patients receive Peacefully's web-based tool to help with end-of-life planning on day 7.

Group II (control): Patients receive standard of care.

After completion of study, patients are followed up at 4, 12, and 24 weeks post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of poor prognosis advanced cancer defined as locally advanced or metastatic cancer and/or disease progression following at least first line systemic therapy
* Access to a computer or mobile device
* The ability to provide informed consent

Exclusion Criteria:

* Not fluent in English
* Severely cognitively impaired (as measured by Short Portable Mental Status Questionnaire scores of < 6)
* Too ill or weak to complete the interviews (as judged by the interviewer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Accrual | Up to 36 months
  The number of participants enrolled during the recruitment period.
Retention rates | Up to 36 months
  The number of participants who completed all study activities.
Change in patients' engagement in advance care planning, as measured by the Decision Maker subscale of the Advance Care Planning Engagement Survey: Action Measures, from baseline to 4 weeks post-randomization | Baseline and Week 4 post-randomization
  Change in patient engagement in advance care planning will be assessed in patients using the reliable and valid Decision Maker (four items) subscale of the Advance Care Planning Engagement Survey: Action Measures. Response options include: yes=1, no=0. Questions include those asking about whether patients have engaged in a decision around advance care planning (e.g., "Have you already decided who you want your medical decision maker to be?" Individual scores can range from 0 to 4, with higher scores indicating that more decisions have been made around advance care planning. Change scores can range from -4 to +4.
Change in patients' engagement in advance care planning, as measured by the Decision Maker subscale of the Advance Care Planning Engagement Survey: Action Measures, from baseline to 12 weeks post-randomization | Baseline and Week 12 post-randomization
  Change in patient engagement in advance care planning will be assessed in patients using the reliable and valid Decision Maker (four items) subscale of the Advance Care Planning Engagement Survey: Action Measures. Response options include: yes=1, no=0. Questions include those asking about whether patients have engaged in a decision around advance care planning (e.g., "Have you already decided who you want your medical decision maker to be?" Individual scores can range from 0 to 4, with higher scores indicating that more decisions have been made around advance care planning. Change scores can range from -4 to +4.
Change in patients' engagement in advance care planning, as measured by the Decision Maker subscale of the Advance Care Planning Engagement Survey: Action Measures, from baseline to 24 weeks post-randomization | Baseline and Week 24 post-randomization
  Change in patient engagement in advance care planning will be assessed in patients using the reliable and valid Decision Maker (four items) subscale of the Advance Care Planning Engagement Survey: Action Measures. Response options include: yes=1, no=0. Questions include those asking about whether patients have engaged in a decision around advance care planning (e.g., "Have you already decided who you want your medical decision maker to be?" Individual scores can range from 0 to 4, with higher scores indicating that more decisions have been made around advance care planning. Change scores can range from -4 to +4.
Change in patients' engagement in advance care planning, as measured by the Quality of Life subscale of the Advance Care Planning Engagement Survey: Action Measures, from baseline to 4 weeks post-randomization | Baseline and Week 4 post-randomization
  Change in patient engagement in advance care planning will be assessed in patients using the reliable and valid Quality of Life (four items) subscale of the Advance Care Planning Engagement Survey: Action Measures. Response options include: yes=1, no=0. Questions include those asking about whether patients have engaged in a decision around quality of life in advance care planning (e.g., "Have you already decided whether or not certain health situations would make your life not worth living?" Individual scores can range from 0 to 4, with higher scores indicating that more decisions have been made around advance care planning as it pertains to quality of life. Change scores can range from -4 to +4.
Change in patients' engagement in advance care planning, as measured by the Quality of Life subscale of the Advance Care Planning Engagement Survey: Action Measures, from baseline to 12 weeks post-randomization | Baseline and Week 12 post-randomization
  Change in patient engagement in advance care planning will be assessed in patients using the reliable and valid Quality of Life (four items) subscale of the Advance Care Planning Engagement Survey: Action Measures. Response options include: yes=1, no=0. Questions include those asking about whether patients have engaged in a decision around quality of life in advance care planning (e.g., "Have you already decided whether or not certain health situations would make your life not worth living?" Individual scores can range from 0 to 4, with higher scores indicating that more decisions have been made around advance care planning as it pertains to quality of life. Change scores can range from -4 to +4.
Change in patients' engagement in advance care planning, as measured by the Quality of Life subscale of the Advance Care Planning Engagement Survey: Action Measures, from baseline to 24 weeks post-randomization | Baseline and Week 24 post-randomization
  Change in patient engagement in advance care planning will be assessed in patients using the reliable and valid Quality of Life (four items) subscale of the Advance Care Planning Engagement Survey: Action Measures. Response options include: yes=1, no=0. Questions include those asking about whether patients have engaged in a decision around quality of life in advance care planning (e.g., "Have you already decided whether or not certain health situations would make your life not worth living?" Individual scores can range from 0 to 4, with higher scores indicating that more decisions have been made around advance care planning as it pertains to quality of life. Change scores can range from -4 to +4.
Change in advance care planning engagement: conversations discussing EoL care, living will, HCP, and DNR orders with family members and loved ones, from baseline to 4 weeks post-randomization | Baseline and Week 4 post-randomization
  Engagement in ACP with family members and loved ones will be assessed in patients. This outcome will consist of documentation of ACP conversations using the investigators' previously utilized 8-item measure of discussing EoL care, living will, HCP, and DNR orders with family (4 items) and doctors (4 items). Scores for the family subscale are computed by summing together the total number of ACP topic discussed with the patient's family members and loved ones. Scores can range from 0 to 4, with higher scores indicating increases in engagement in ACP conversations with family members and loved ones.
Change in advance care planning engagement: conversations discussing EoL care, living will, HCP, and DNR orders with family members and loved ones, from baseline to 12 weeks post-randomization | Baseline and Week 12 post-randomization
  Engagement in ACP with family members and loved ones will be assessed in patients. This outcome will consist of documentation of ACP conversations using the investigators' previously utilized 8-item measure of discussing EoL care, living will, HCP, and DNR orders with family (4 items) and doctors (4 items). Scores for the family subscale are computed by summing together the total number of ACP topic discussed with the patient's family members and loved ones. Scores can range from 0 to 4, with higher scores indicating increases in engagement in ACP conversations with family members and loved ones.
Change in advance care planning engagement: conversations discussing EoL care, living will, HCP, and DNR orders with family members and loved ones, from baseline to 24 weeks post-randomization | Baseline and Week 24 post-randomization
  Engagement in ACP with family members and loved ones will be assessed in patients. This outcome will consist of documentation of ACP conversations using the investigators' previously utilized 8-item measure of discussing EoL care, living will, HCP, and DNR orders with family (4 items) and doctors (4 items). Scores for the family subscale are computed by summing together the total number of ACP topic discussed with the patient's family members and loved ones. Scores can range from 0 to 4, with higher scores indicating increases in engagement in ACP conversations with family members and loved ones.
Change in advance care planning engagement: conversations discussing EoL care, living will, HCP, and DNR orders with doctors, from baseline to 4 weeks post-randomization | Baseline and Week 4 post-randomization
  Engagement in ACP with doctors will be assessed in patients. This outcome will consist of documentation of ACP conversations using the investigators' previously utilized 8-item measure of discussing EoL care, living will, HCP, and DNR orders with family (4 items) and doctors (4 items). Scores for the doctor subscale are computed by summing together the total number of ACP topic discussed with the patient's doctors. Scores can range from 0 to 4, with higher scores indicating increases in engagement in ACP conversations with doctors.
Change in advance care planning engagement: conversations discussing EoL care, living will, HCP, and DNR orders with doctors, from baseline to 12 weeks post-randomization | Baseline and Week 12 post-randomization
  Engagement in ACP with doctors will be assessed in patients. This outcome will consist of documentation of ACP conversations using the investigators' previously utilized 8-item measure of discussing EoL care, living will, HCP, and DNR orders with family (4 items) and doctors (4 items). Scores for the doctor subscale are computed by summing together the total number of ACP topic discussed with the patient's doctors. Scores can range from 0 to 4, with higher scores indicating increases in engagement in ACP conversations with doctors.
Change in advance care planning engagement: conversations discussing EoL care, living will, HCP, and DNR orders with doctors, from baseline to 24 weeks post-randomization | Baseline and Week 24 post-randomization
  Engagement in ACP with doctors will be assessed in patients. This outcome will consist of documentation of ACP conversations using the investigators' previously utilized 8-item measure of discussing EoL care, living will, HCP, and DNR orders with family (4 items) and doctors (4 items). Scores for the doctor subscale are computed by summing together the total number of ACP topic discussed with the patient's doctors. Scores can range from 0 to 4, with higher scores indicating increases in engagement in ACP conversations with doctors.
Change in advance care planning engagement: completion of advance directives, from baseline to 4 weeks post-randomization | Baseline and Week 4 post-randomization
  Completion of advance directives will be assessed by asking patients whether they completed a do-not-resuscitate order, a living will, and/or identified a health care proxy; data will be verified through the patient's electronic health record. Change in these numbers will be assessed at baseline and post-intervention. Scores are computed by summing together the total number of advance directives completed. Scores can range from 0 to 3, with higher scores indicating increases in completion of advance directives. Change scores can range from -3 to +3.
Change in advance care planning engagement: completion of advance directives, from baseline to 12 weeks post-randomization | Baseline and Week 12 post-randomization
  Completion of advance directives will be assessed by asking patients whether they completed a do-not-resuscitate order, a living will, and/or identified a health care proxy; data will be verified through the patient's electronic health record. Change in these numbers will be assessed at baseline and post-intervention. Scores are computed by summing together the total number of advance directives completed. Scores can range from 0 to 3, with higher scores indicating increases in completion of advance directives. Change scores can range from -3 to +3.
Change in advance care planning engagement: completion of advance directives, from baseline to 24 weeks post-randomization | Baseline and Week 24 post-randomization
  Completion of advance directives will be assessed by asking patients whether they completed a do-not-resuscitate order, a living will, and/or identified a health care proxy; data will be verified through the patient's electronic health record. Change in these numbers will be assessed at baseline and post-intervention. Scores are computed by summing together the total number of advance directives completed. Scores can range from 0 to 3, with higher scores indicating increases in completion of advance directives. Change scores can range from -3 to +3.

SECONDARY OUTCOMES:
Change in comprehensive end-of-life planning, from baseline to 4 weeks post-randomization | Baseline and Week 4 post-randomization
  Will be measured using a 15-item checklist of all completed tasks from the checklists/tasks on the website (eg, gather important documents, create a will). Scores are computed by summing together the total number of planning items completed. Scores can range from 0 to 15, with higher scores indicating increases in completion of end-of-life planning tasks. Change scores can range from -15 to +15.
Change in comprehensive end-of-life planning, from baseline to 12 weeks post-randomization | Baseline and Week 12 post-randomization
  Will be measured using a 15-item checklist of all completed tasks from the checklists/tasks on the website (eg, gather important documents, create a will). Scores are computed by summing together the total number of planning items completed. Scores can range from 0 to 15, with higher scores indicating increases in completion of end-of-life planning tasks. Change scores can range from -15 to +15.
Change in comprehensive end-of-life planning, from baseline to 24 weeks post-randomization | Baseline and Week 24 post-randomization
  Will be measured using a 15-item checklist of all completed tasks from the checklists/tasks on the website (eg, gather important documents, create a will). Scores are computed by summing together the total number of planning items completed. Scores can range from 0 to 15, with higher scores indicating increases in completion of end-of-life planning tasks. Change scores can range from -15 to +15.
Change in psychological distress, as measured by the Hospital Anxiety and Depression Scale (HADS), from baseline to 4 weeks post-randomization | Baseline and Week 4 post-randomization
  Psychological distress will be measured using the Hospital Anxiety and Depression Scale (HADS), a valid and reliable 14-item, Likert-type self-report measure of mood disturbance commonly used with cancer patients. The HADS contains two seven-item subscales: 1) anxiety and 2) depressive symptoms. Each item on this scale is rated on a 4-point scale (0 to 3), and all items are summed to create a HADS total score. Total scores can range from 0 to 42, with higher numbers indicating higher levels of distress. Change in psychological distress will be assessed at baseline and post-randomization.
Change in psychological distress, as measured by the Hospital Anxiety and Depression Scale (HADS), from baseline to 12 weeks post-randomization | Baseline and Week 12 post-randomization
  Psychological distress will be measured using the Hospital Anxiety and Depression Scale (HADS), a valid and reliable 14-item, Likert-type self-report measure of mood disturbance commonly used with cancer patients. The HADS contains two seven-item subscales: 1) anxiety and 2) depressive symptoms. Each item on this scale is rated on a 4-point scale (0 to 3), and all items are summed to create a HADS total score. Total scores can range from 0 to 42, with higher numbers indicating higher levels of distress. Change in psychological distress will be assessed at baseline and post-randomization.
Change in psychological distress, as measured by the Hospital Anxiety and Depression Scale (HADS), from baseline to 24 weeks post-randomization | Baseline and Week 24 post-randomization
  Psychological distress will be measured using the Hospital Anxiety and Depression Scale (HADS), a valid and reliable 14-item, Likert-type self-report measure of mood disturbance commonly used with cancer patients. The HADS contains two seven-item subscales: 1) anxiety and 2) depressive symptoms. Each item on this scale is rated on a 4-point scale (0 to 3), and all items are summed to create a HADS total score. Total scores can range from 0 to 42, with higher numbers indicating higher levels of distress. Change in psychological distress will be assessed at baseline and post-randomization.
Change in emotional well-being, as measured by the Functional Assessment of Cancer Therapy-General (FACT-G) scale, from baseline to 4 weeks post-randomization | Baseline and Week 4 post-randomization
  Emotional well-being will be measured using the emotional well-being subscale of the 27-item Functional Assessment of Cancer Therapy-General (FACT-G) scale. The FACT-G scale contains 27 items, of which 6 measure emotional well-being. Items on the FACT-G ask patients to rate the degree to which they agree to statements about their well-being. Each item on this scale is rated on a 5-point Likert scale (1 = not at all, 5 = very much), with higher scores indicating better well-being. Total scores for the emotional well-being subscale can range from 6 to 30. Change in emotional well-being will be assessed at baseline and 4 weeks post-randomization.
Change in emotional well-being, as measured by the Functional Assessment of Cancer Therapy-General (FACT-G) scale, from baseline to 12 weeks post-randomization | Baseline and Week 12 post-randomization
  Emotional well-being will be measured using the emotional well-being subscale of the 27-item Functional Assessment of Cancer Therapy-General (FACT-G) scale. The FACT-G scale contains 27 items, of which 6 measure emotional well-being. Items on the FACT-G ask patients to rate the degree to which they agree to statements about their well-being. Each item on this scale is rated on a 5-point Likert scale (1 = not at all, 5 = very much), with higher scores indicating better well-being. Total scores for the emotional well-being subscale can range from 6 to 30. Change in emotional well-being will be assessed at baseline and 4 weeks post-randomization.
Change in emotional well-being, as measured by the Functional Assessment of Cancer Therapy-General (FACT-G) scale, from baseline to 24 weeks post-randomization | Baseline and Week 24 post-randomization
  Emotional well-being will be measured using the emotional well-being subscale of the 27-item Functional Assessment of Cancer Therapy-General (FACT-G) scale. The FACT-G scale contains 27 items, of which 6 measure emotional well-being. Items on the FACT-G ask patients to rate the degree to which they agree to statements about their well-being. Each item on this scale is rated on a 5-point Likert scale (1 = not at all, 5 = very much), with higher scores indicating better well-being. Total scores for the emotional well-being subscale can range from 6 to 30. Change in emotional well-being will be assessed at baseline and 4 weeks post-randomization.
Change in social/family well-being, as measured by the Functional Assessment of Cancer Therapy-General scale, from baseline to 4 weeks post-randomization | Baseline and Week 4 post-randomization
  Social well-being will be measured using the social well-being subscale of the 27-item Functional Assessment of Cancer Therapy-General (FACT-G) scale. The FACT-G scale contains 27 items, of which 7 measure social/family well-being. Items on the FACT-G ask patients to rate the degree to which they agree to statements about their well-being. Each item on this scale is rated on a 5-point Likert scale (1 = not at all, 5 = very much), with higher scores indicating better well-being. Total scores for the social/family well-being subscale can range from 6 to 35. Change in social/family well-being will be assessed at baseline and 4 weeks post-randomization.
Change in social/family well-being, as measured by the Functional Assessment of Cancer Therapy-General scale, from baseline to 12 weeks post-randomization | Baseline and Week 12 post-randomization
  Social well-being will be measured using the social well-being subscale of the 27-item Functional Assessment of Cancer Therapy-General (FACT-G) scale. The FACT-G scale contains 27 items, of which 7 measure social/family well-being. Items on the FACT-G ask patients to rate the degree to which they agree to statements about their well-being. Each item on this scale is rated on a 5-point Likert scale (1 = not at all, 5 = very much), with higher scores indicating better well-being. Total scores for the social/family well-being subscale can range from 6 to 35. Change in social/family well-being will be assessed at baseline and 4 weeks post-randomization.
Change in social/family well-being, as measured by the Functional Assessment of Cancer Therapy-General scale, from baseline to 24 weeks post-randomization | Baseline and Week 24 post-randomization
  Social well-being will be measured using the social well-being subscale of the 27-item Functional Assessment of Cancer Therapy-General (FACT-G) scale. The FACT-G scale contains 27 items, of which 7 measure social/family well-being. Items on the FACT-G ask patients to rate the degree to which they agree to statements about their well-being. Each item on this scale is rated on a 5-point Likert scale (1 = not at all, 5 = very much), with higher scores indicating better well-being. Total scores for the social/family well-being subscale can range from 6 to 35. Change in social/family well-being will be assessed at baseline and 4 weeks post-randomization.
Change in spiritual well-being, as measured by the Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being Scale (FACIT-Sp), from baseline to 4 weeks post-randomization | Baseline and Week 4 post-randomization
  Spiritual well-being will be measured using the validated, 12-item Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being Scale (FACIT-Sp). The FACIT-Sp asks patients to indicate the degree to which they agree with statements about their spiritual well-being. Each item on this scale is rated on a 5-point Likert scale (0 = not at all, 4 = very much), with higher scores indicating greater spiritual well-being. Total scores range from 0 to 48. Change in spiritual well-being will be assessed at baseline and 4 weeks post-randomization.
Change in spiritual well-being, as measured by the Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being Scale, from baseline to 12 weeks post-randomization | Baseline and Week 12 post-randomization
  Spiritual well-being will be measured using the validated, 12-item Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being Scale (FACIT-Sp). The FACIT-Sp asks patients to indicate the degree to which they agree with statements about their spiritual well-being. Each item on this scale is rated on a 5-point Likert scale (0 = not at all, 4 = very much), with higher scores indicating greater spiritual well-being. Total scores range from 0 to 48. Change in spiritual well-being will be assessed at baseline and 4 weeks post-randomization.
Change in spiritual well-being, as measured by the Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being Scale, from baseline to 24 weeks post-randomization | Baseline and Week 24 post-randomization
  Spiritual well-being will be measured using the validated, 12-item Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being Scale (FACIT-Sp). The FACIT-Sp asks patients to indicate the degree to which they agree with statements about their spiritual well-being. Each item on this scale is rated on a 5-point Likert scale (0 = not at all, 4 = very much), with higher scores indicating greater spiritual well-being. Total scores range from 0 to 48. Change in spiritual well-being will be assessed at baseline and 4 weeks post-randomization.
Change in financial well-being, as measured by the InCharge Financial Distress/Financial Well-Being scale, from baseline to 4 weeks post-randomization | Baseline and Week 4 post-randomization
  Financial well-being will be measured using the validated, 8-item InCharge Financial Distress/Financial Well-Being scale. This scale asks patients to rate their financial wellness (stress, satisfaction, etc.) on a 10-point Likert scale that varies for each response but for which 1 indicates the lowest financial well-being and 10 indicates the highest (e.g., 1=overwhelming stress to 10 = not stress at all; 1 = worry all the time, 10 - never worry). Total scores range from 8 to 80, with higher scores indicating greater financial well-being. Change in financial well-being will be assessed at baseline and 4 weeks post-randomization.
Change in financial well-being, as measured by the InCharge Financial Distress/Financial Well-Being scale, from baseline to 12 weeks post-randomization | Baseline and Week 12 post-randomization
  Financial well-being will be measured using the validated, 8-item InCharge Financial Distress/Financial Well-Being scale. This scale asks patients to rate their financial wellness (stress, satisfaction, etc.) on a 10-point Likert scale that varies for each response but for which 1 indicates the lowest financial well-being and 10 indicates the highest (e.g., 1=overwhelming stress to 10 = not stress at all; 1 = worry all the time, 10 - never worry). Total scores range from 8 to 80, with higher scores indicating greater financial well-being. Change in financial well-being will be assessed at baseline and 4 weeks post-randomization.
Change in financial well-being, as measured by the InCharge Financial Distress/Financial Well-Being scale, from baseline to 24 weeks post-randomization | Baseline and Week 24 post-randomization
  Financial well-being will be measured using the validated, 8-item InCharge Financial Distress/Financial Well-Being scale. This scale asks patients to rate their financial wellness (stress, satisfaction, etc.) on a 10-point Likert scale that varies for each response but for which 1 indicates the lowest financial well-being and 10 indicates the highest (e.g., 1=overwhelming stress to 10 = not stress at all; 1 = worry all the time, 10 - never worry). Total scores range from 8 to 80, with higher scores indicating greater financial well-being. Change in financial well-being will be assessed at baseline and 4 weeks post-randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Megan J. Shen, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT05564468/ICF_000.pdf